CLINICAL TRIAL: NCT07405684
Title: Clinical Efficacy and Health Economic Evaluation of Fecal Molecular Susceptibility-guided Therapy for Helicobacter Pylori Infection First-line Treatment: Multicenter Randomized Controlled Study
Brief Title: Fecal Molecular Susceptibility-guided Hp First-line Therapy
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B2026-013-1
Record Dates: First submitted 2026-02-05; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: HELICOBACTER PYLORI INFECTIONS
Keywords: Helicobacter pylori

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 7-day (Experimental)
  Interventions: Drug: 7-day fecal molecular susceptibility-guided therapy
- 14-day (Active Comparator)
  Interventions: Drug: 14-day fecal molecular susceptibility-guided therapy

INTERVENTIONS:
Drug: 7-day fecal molecular susceptibility-guided therapy — This intervention involves performing polymerase chain reaction (PCR)-based detection of Helicobacter pylori drug resistance genes (including clarithromycin, levofloxacin) from fecal samples. Based on the susceptibility results and penicillin-allergic test, a tailored 7-day triple or quadruple therapy regimen is prescribed, including Tegoprazan , Amoxicillin, Clarithromycin, Levofloxacin, Bismuth Potassium Citrate, Metronidazole, Doxycycline or Minocycline.
  Arms: 7-day
Drug: 14-day fecal molecular susceptibility-guided therapy — This intervention involves performing polymerase chain reaction (PCR)-based detection of Helicobacter pylori drug resistance genes (including clarithromycin, levofloxacin) from fecal samples. Based on the susceptibility results, a tailored 14-day triple or quadruple therapy regimen is prescribed, including Tegoprazan , Amoxicillin, Clarithromycin, Levofloxacin, Bismuth Potassium Citrate, Metronidazole, Doxycycline or Minocycline.
  Arms: 14-day

SUMMARY:
The goal of this clinical trial is to evaluate the eradication efficacy and health economic benefits of individualized regimens guided by fecal molecular susceptibility testing with 7-day and 14-day courses in the first-line treatment of Helicobacter pylori infection. The main questions it aims to answer are:

1. What is the H. pylori eradication rate of the 7-day versus 14-day individualized regimens?
2. What are the safety, adherence, and cost-effectiveness of the 7-day versus 14-day individualized regimens? Researchers will compare the 7-day course group and the 14-day course group to see if the 7-day course is non-inferior to the 14-day course in terms of eradication rate.

Participants will:

1. Undergo fecal H. pylori drug resistance gene testing
2. Receive randomized assignment to either 7-day or 14-day individualized treatment based on drug susceptibility results
3. Complete follow-up visits at 1 week and 4-8 weeks after stopping treatment for adverse event monitoring and 13C-urea breath test

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in this clinical study; fully understand, be informed about this study, and sign the Informed Consent Form (ICF).
2. Age between 18 and 75 years (inclusive) on the day of signing the ICF.
3. 13C-urea breath test (13C-UBT) and fecal HP nucleic acid detection confirming Helicobacter pylori (Hp) infection.
4. Not previously eradicated HP

Exclusion Criteria:

1. Individuals with a known allergy to the medication.
2. Patients with severe cardiovascular, pulmonary, renal, hepatic, hematologic, neurologic, endocrine, or psychiatric disorders;
3. Participants or guardians who refuse to enroll;
4. Alcohol and/or drug abuse (dependence or addiction) or individuals judged by the physician to have poor compliance; 5) Use of antibiotics, bismuth-containing drugs, PPIs, or traditional Chinese medicines within 4 weeks before treatment; 6) Pregnant or lactating women; 7) Any condition deemed by the investigator to be unsuitable for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 544 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Eradication rate of Helicobacter pylori | 4-8 weeks after treatment
  Eradication of Helicobacter pylori was defined as negative result of urea breath test (<4‰ cut-off value)

SECONDARY OUTCOMES:
Frequency of adverse events | Throughout the treatment period, up to 2 weeks
  Any possible adverse events during the treatment period were recorded.
Adherence rate | Throughout the treatment period, up to 2 weeks
  The proportion of subjects with good adherence. Good adherence was defined as that subjects took more than 80% of the total medication.

OTHER OUTCOMES:
Average cost of each group | Throughout the treatment period, up to 2 weeks
  Average medical cost related to therapy and followup in each group

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Renji Hospital, School of Medicine, Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - Shanghai Jiangong Hospitail., Shanghai, Shanghai Municipality
  - Shanghai Tenth People Hospital, Shanghai, Shanghai Municipality
  - Zhongshan Hospital, Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: No